CLINICAL TRIAL: NCT02426034
Title: Safety and Efficacy of Apatinib in Patients With Advanced Gastric or Gastroesophageal Junction Adenocarcinoma After Failure of Two or More Lines of Chemotherapy (Ahead-G201): a Prospective, Single-arm, Multicenter, Phase IV Study
Brief Title: A Study of Apatinib Tablets in the Treatment of Advanced or Metastatic Gastric Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ahead-G201
Record Dates: First submitted 2015-04-09; First posted 2015-04-24 (Estimated); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Advanced Gastric or Gastroesophageal Junction Adenocarcinoma
Keywords: Advanced; Metastatic
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: A large-scale single-arm phase IV study

ARMS (1):
- Treatment group (Experimental): Apatinib Tablets
  Interventions: Drug: ApatinibTablets

INTERVENTIONS:
Drug: ApatinibTablets — Apatinib Tablets, recommended dose of 850mg

SUMMARY:
The large-scale phase IV study aims to verify the safety and efficacy of apatinib in patients with advanced gastric cancer or gastroesophageal junction adenocarcinoma after failure of two lines of chemotherapy. Apatinib initiated at a recommended dose of 850mg. However, the starting dose was decided by investigator's choice based on patients' condition. Dose interruption and dose reduction were allowed according to the product label. Treatment continued until disease progression, intolerable toxicity, withdrawal of informed consent, or at investigators' discretion. The primary endpoint was safety, which was assessed by recording the incidence and severity of adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to75 years old;
2. Pathologically diagnosed with advanced gastric cancer (including adenocarcinoma of the gastroesophageal junction);
3. Failure of prior therapy (during or after treatment) in patients who have received at least two prior chemotherapy regimens;
4. ECOG PS of 0-2;
5. Major organ function has to meet the following criteria:

   For results of blood routine test (without blood transfusion within 14 days):

   HB ≥ 90g / L ANC ≥ 1.5 × 109 / L PLT ≥ 80 × 109 / L

   Biochemical tests results:

   Bilirubin <1.25 times the upper limit of normal (ULN) ALT and AST <2.5 × ULN; liver metastases, if any, the ALT and AST<5 × ULN Serum Cr ≤ 1 × ULN endogenous creatinine clearance>50ml/min (Cockcroft-Gault formula)
6. An expected survival of ≥ 3 months;
7. Patient received apatinib treatment regimen at investigators' discretion;
8. Patient has to voluntarily join the study and sign the Informed Consent Form for the study;
9. Pregnancy test (serum or urine) has to be performed for woman of childbearing age within 7 days before enrolment and the test result must be negative. They shall take appropriate methods for contraception during the study until the 8th week post the last administration of study drug. For men, (previous surgical sterilization accepted), shall agree to take appropriate methods of contraception during the study until the 8th week post the last administration of study drug.

Exclusion Criteria:

1. Subjects with uncontrolled arterial hypertension (systolic blood pressure> 140 mmHg and diastolic blood pressure > 90 mm Hg) despite standard medical management; Grade ≥ 2 coronary heart disease; Grade ≥ 2 arrhythmia (including QT interval prolongation, for man > 450 ms, for woman > 470 ms), as well as Grade ≥ 2 cardiac dysfunction;
2. Factors that could have an effect on oral medication (such as inability to swallow, chronic diarrhea and intestinal obstruction);
3. Subjects with high gastrointestinal bleeding risk, including the following conditions: presence of active ulceration combined with a positive fecal occult blood test (++);history of hematemesis and melena within three months before enrollment; unresected primary lesion in stomach with positive fecal occult blood test (+), ulcerated gastric carcinoma with massive alimentary tract bleeding risk judged by PIs based on gastric endoscopy finding;
4. Abnormal coagulation (INR>1.5、APTT>1.5 UNL), with tendency of bleeding;
5. Presence of central nervous system metastases;
6. Pregnant or lactating women;
7. Other conditions regimented at investigators' discretion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2004 (Actual)
Dates: Start 2015-05-15 (Actual); Primary Completion 2020-05-29 (Actual); Study Completion 2020-09-03 (Actual)

PRIMARY OUTCOMES:
Safety, which was assessed by recording the incidence and severity of adverse events | between first dose of apatinib and up to 30 days after the last dose of apatinib

SECONDARY OUTCOMES:
Overall Survival | Event driven, an expected average of 34 weeks
Progression Free Survival | An expected average of 12 weeks
Objective Response Rate | An expected average of 12 weeks
Disease Control Rate | An expected average of 12 weeks
Quality of life, measured by the questionnaire of EORTC QLQ-C30 | Quality of life will be assessed at baseline (after the patients provided written informed consent) until at least 4 weeks after the last dose of study drug was administered, an expected average of 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, MD, Principal Investigator — Fudan University
Locations (2):
- China (2):
  - Nanjin Military 81 Hosiptal, Nanjing, Jiangsu
  - Fudan University cancer hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li J, Qin S, Wen L, Wang J, Deng W, Guo W, Jia T, Jiang D, Zhang G, He Y, Ba Y, Zhong H, Wang L, Lin X, Yang J, Zhao J, Bai Y, Wu X, Gao F, Sun G, Wu Y, Ye F, Wang Q, Xie Z, Yi T, Huang Y, Yu G, Lu L, Yuan Y, Li W, Liu L, Sun Y, Sun Y, Yin L, Hou Z. Safety and efficacy of apatinib in patients with advanced gastric or gastroesophageal junction adenocarcinoma after the failure of two or more lines of chemotherapy (AHEAD): a prospective, single-arm, multicenter, phase IV study. BMC Med. 2023 May 5;21(1):173. doi: 10.1186/s12916-023-02841-7. PMID 37147645